CLINICAL TRIAL: NCT06524856
Title: The Increase of Lung Capacity Using the Lung Master (Pulmonary Exerciser)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0108-24-EP
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Dyspnea; Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Intervention Model Description: The Lung Master will force the lung muscle to work more strenuously and gradually build breathing muscles. Therefore, this study will focus on determining how The Lung Master (Pulmonary Exerciser) increases lung capacity in healthy participants, which leads to improved overall lung functioning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Function in Young and Older Adults (Experimental): Lung functions will be assess for two groups: young and older adults. The age range of 19 to 35 is categorized as young adulthood. This age range was selected because the lungs mature around 19-25 years old. The age range above 65 is designated as late adulthood, where lung function gradually declines.
  Interventions: Device: Lung Master (Pulmonary Exerciser)

INTERVENTIONS:
Device: Lung Master (Pulmonary Exerciser) — During the one-month using the Lung Master at their house, the participant will be using it at least one time every day, either in the morning or in the evening before going to sleep. During the session, the participants will sit upright and try to prolong the inhalation and exhalation breaths through the Lung Master device for at least three seconds. For each session, the participants will try to concentrate on 35-50 breaths in and breaths out which is about 2-5 minutes. Every session can involve using the Pulmonary Exerciser for a minimum of 5 minutes and a maximum of 20 minutes. After each session, participants will be asked to note how long they have used the device and when they have used it. Information from each session will be recorded on the Participant Device Log that will be provided.

SUMMARY:
Investigators are studying how a device called The Lung Master device can help people breathe better. The investigational device increases the amount of air our lungs can hold, which is important for overall lung health. The Lung Master is not approved by the FDA.

The study has two visits approximately one month apart. In the first visit participants will take a spirometry test, particularly forced vital capacity (FVC), to measure volume change in the lungs. Participants will take the investigational device home to use daily, either in the morning or evening. Use will be recorded in a diary. After one month, participants will return for another spirometry test. Each study visit will take about one to two hours to complete.

DETAILED DESCRIPTION:
Shortness of breath,or dyspnea, occurs when the lungs do not receive enough oxygen leading to discomfort when breathing. This occurs in a quarter of individuals seen in an outpatient setting. Several factors can relate to breathlessness, including lung disorders, heart conditions, or stress. Patients with breathlessness often experience physical limitations in their daily activities. Various treatments for dyspnea are available, however, chronic breathlessness syndrome, such as asthma or chronic obstructive pulmonary disease (COPD), still can persist even when treatment is available.

The Lung Master (Pulmonary Exerciser) is a breathing device used for the respiratory treatment and rehabilitation of chronic breathlessness syndrome. The Lung Master increases resistance during inhalation and exhalation, which works to strengthen the respiratory muscle and improve overall lung function. Therefore, this study will focus on determining how the Lung Master increases lung capacity in healthy individuals. The device is considered investigational and has not been approved by the FDA.

Two groups of healthy participants will be sought for the study: ages 19 to 35 and ages 65 and above. Each participant will have two in-office study visits approximately one month apart. Each visit will take around one to two hours to complete. At the visits, a breathing test called a spirometry test will be done. During the one month interim, the study device will be used at home and the use recorded in a diary. The device must be used least once every day, either in the morning or in the evening for 5 to 20 minutes. You will be contacted after two weeks, and then return the device at the second study visit.

ELIGIBILITY:
Inclusion Criteria:

* able to complete the at home portion of the study daily
* fall within the age ranges: 19-35 and above 65 years old

Exclusion Criteria:

* any respiratory or chronic conditions

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Inspiratory Capacity | baseline and after one month of device use
  After reaching the end of a normal, quiet expiration, the maximum volume of air that can be inspired will be measured.
Tidal Volume | baseline and after one month of device use
  The amount of air that moves in or out of the lungs with each respiratory cycle will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Farahnaz Fallah Tafti, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Biomechanics Research Building, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berliner D, Schneider N, Welte T, Bauersachs J. The Differential Diagnosis of Dyspnea. Dtsch Arztebl Int. 2016 Dec 9;113(49):834-845. doi: 10.3238/arztebl.2016.0834. PMID 28098068
- [Background] Sandberg J, Olsson M, Ekstrom M. Underlying conditions contributing to breathlessness in the population. Curr Opin Support Palliat Care. 2021 Dec 1;15(4):219-225. doi: 10.1097/SPC.0000000000000568. PMID 34610625
- [Background] David S, Goldin J, Edwards CW. Forced Expiratory Volume. 2024 Oct 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK540970/ PMID 31082014
- [Background] Nguyen JD, Duong H. Pursed-lip Breathing. 2025 Jan 25. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK545289/ PMID 31424873